CLINICAL TRIAL: NCT04531228
Title: Sun Yat-sen University Cancer Center
Brief Title: TACE-HAIC Plus Lenvatinib for Patients With Unresectable HCC: an Open-label, Single-arm, Phase 2 Trial
Acronym: Thalen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yunfei Yuan (Other)
Responsible Party: Sponsor-Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-137
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma; Transarterial Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: TACE-HAIC plus lenvatinib (Experimental): chemo-lipiodolization, followed by FOLFOX-based chemotherapy artery infusion (HAIC). Lenvatinib was administrated two or four days after TACE-HAIC.
  Interventions: Procedure: TACE-HAIC plus lenvatinib

INTERVENTIONS:
Procedure: TACE-HAIC plus lenvatinib — chemo-lipiodolization with EADM (30mg/m2), followed by FOLFOX-based chemotherapy artery infusion (Oxa 85mg/m2, 5-Fu 400 mg/m2, 5-Fu 1200mg/m2). Lenvatinib was administrated two or four days after TACE-HAIC, with 8mg for patients weight <60kg, or 12mg for patients weight more than 60Kg.

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most commonly malignant tumors around the world. Hepatic resection or liver transplantation is the radical method to cure the disease. However, due to multiple tumors or poor hepatic function reserve in cirrhosis, surgical treatment is suitable for early-stage and well reserved liver function patients. Therefore, in clinical practice, transarterial chemoembolization (TACE) is a preferential and standard treatment of unresectable HCC. TACE has been proved to provide outstanding efficacy for treating advanced stage HCC patients. However, TACE is associated with a high rate of treatment failure for advanced HCC patients. EACH trial opened the door to FOLFOX-based system chemotherapy for advanced HCC patients. Recently, investigators have showed that hepatic arterial infusion of FOLFOX-based chemotherapy (HAIC) was safe and efficient for advanced HCC patients. The combination of TACE with HAIC (TACE-HAIC) was proved to increase the local doses of chemotherapeutic agents in the liver, reduce the viability of HCC cells and increase the hepatectomy rate in our previous study.

Levatinib is a new treatment and offers relative high overall response rate for advanced HCC, which was approved in China and Japan. However, whether the combination of TACE-HAIC and Lenvatinib would increse tumor control for unresectable patients is still unknown. Thus, this single arm, phase 2 study is designed to analyze the safety and efficacy TACE-HAIC plus Lenvatinib for patients with unresectalbe HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years

  1. The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
  2. unresectable disease, stage BCLC B/C
  3. No previous anti-HCC treatment
  4. Eastern Co-operative Group performance status 2 or less
  5. Liver function: Child's A or B (score < 7)

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy

  1. underlying serve cardiac or renal diseases
  2. Known or suspected allergy to the investigational agent or any agent given in association with this trial
  3. Patients ineligible for hepatic artery embolization

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6-12 months
  the time from assignment to progression, death or last follow-up.

SECONDARY OUTCOMES:
overall survival | 6-12 months
  the time from assignment to death or last follow-up
overall response rate | 6-12 months
  Objective response rate defined as confirmed complete response or partial response under mRECIST 1.1 criteria
adverse effects | 6-12 months
  Frequency and severity of adverse effects as defined by CTCAE version 5

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No